CLINICAL TRIAL: NCT03747731
Title: KIDNEY - LUNG INTERACTION: the Effect of End-expiratory Pressure on Renal Perfusion. Non-invasive Evaluation.
Brief Title: A Non-invasive Evaluation of Kidney-Lung Interactions
Acronym: KIDNEY-LUNG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Principal Investigator, Silvia De Rosa, Medical Doctor, St. Bortolo Hospital
Other Study IDs: 88/18
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-11

CONDITIONS: Perfusion; Complications; Mechanical Ventilation Complication
Keywords: Renal blood perfusion; Mechanical ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resistive Index and Peep Titration: Enrolled patients will receive a sequential, step-wise increase in PEEP from 0 cmH2O to 12 cmH2O. The inter-lobar arterioles will be sampled at each PEEP increment and the IR will be measured as the average of three values recorded at the upper and lower pole and at the mesorenes in each kidney.
  Gas exchanges, HR, systolic, diastolic and mean PA, Pmax, P1 and P2 airway, total resistance and ohmic resistance and static respiratory compliance indexed for body weight (RRSmaxI, RRSminI, CrsI) will be measured at each Peep Level.
  The physiologic measurements will be obtained at regular intervals (within 15 minutes at each PEEP level) throughout the PEEP titration period.

SUMMARY:
The present study aims to evaluate, with non-invasive methods, the relationships existing between PEEP and renal perfusion in patients undergoing surgery and requiring ventilatory support and monitoring in intensive care. Renal perfusion will be assessed at baseline (PEEP 0), subsequently ,at the application of progressive increases of PEEP. At the end of the measurements, the implications of the use of PEEP on the renal vascular system will be analyzed.

DETAILED DESCRIPTION:
The present physiological, monocentric, observational clinical study evaluates the effect of progressive PEEP increases on renal perfusion in mechanically ventilated patients who underwent surgery with the need of ventilatory support and monitoring in intensive care.

Precisely, will be evaluated:

* The morphometric parameters (coronal diameter and cortico-medullary thickness) and the renal resistive indices (IR). The inter-lobar arteries will be sampled and the IRs will be measured as the upper and lower level and the mesorenes. Measurements will be performed both in the kidney and in baseline conditions and incremental values of PEEP (0 - 6 - 12).
* Gas exchanges, FC, systolic BP, diastolic and mean, Pmax, P1 and P2 of the airways, total and ohmic resistances and static respiratory compliance indexed for weight body (RRSmaxI, RRSminI, CrsI will be recorded).

The intra-class correlation coefficient will be measured to estimate the intra-observer reproducibility of the conducted measurement.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Receiving mechanical ventilation, invasive blood pressure monitoring and an urinary catheter to monitor diuresis
* Need for postoperative monitoring in intensive care
* Written informed consent;

Exclusion Criteria:

* Acute kidney injury defined according to KDIGO guidelines;
* Pre-existing chronic renal disease;
* Heart failure;
* ARDS;
* Sepsis and Septic Shock;
* Hemodynamic instability with the need for vasoactive support;
* Chronic or occasional therapy with drugs that could modify the renal blood flow and that can not be suspended two days before the study (Vasoactive agents, Ace-inhibitors, Beta-blockers, NSAIDs, Sartans and Diuretics therapy);
* Presumed or established state of pregnancy;
* Refusal of informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery and with the need for ventilatory support for the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-05-19 (Estimated); Study Completion 2019-11-19 (Estimated)

PRIMARY OUTCOMES:
Association between IR and PEEP | Change from baseline to 60 minutes
  Resistive index will be measured in both kidney and recorded using multifrequency convex probe.The association between positive end expiratory pressure and resistive index will be analyzed as the primary outcome.

SECONDARY OUTCOMES:
Association between PEEP and Hemodynamics Paramenters | Change from baseline to 60 minutes
  Resistive index will be measured in both kidney and recorded using multifrequency convex. FC, systolic, diastolic and mean PA will be measured at each PEEP level

OTHER OUTCOMES:
Association between IR and Respiratory exchanges | Change from baseline to 60 minutes
  Resistive index will be measured in both kidney and recorded using multifrequency convex. PaO2 and PaCO2 will be analyzed at each PEEP level.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia De Rosa, MD, Principal Investigator — Ospedale San Bortolo di Vicenza
Locations (1):
- San Bortolo Hospital, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: No